CLINICAL TRIAL: NCT00043394
Title: A Phase I/II Open Label, Multi-Center, Dose-Escalation Study Of Subcutaneous CPG 7909 Plus Herceptin® In Patients With Metastatic Breast Cancer
Brief Title: CPG 7909 Plus Herceptin® In Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C015; A8501021, CO15
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Carcinoma, Breast
Keywords: CpG 7909 subcutaneous injection combination with Herceptin® metastatic breast cancer.
MeSH Terms: conditions — Breast Neoplasms | interventions — ProMune; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 0.04 mg/kg CpG 7909
  Interventions: Drug: 0.04 mg/kg CpG 7909; Drug: Herceptin®
- Cohort 2 (Experimental): 0.08 mg/kg CpG 7909
  Interventions: Drug: 0.08 mg/kg CpG 7909; Drug: Herceptin®
- Cohort 3 (Experimental): 0.12 mg/kg CpG 7909 Injection once weekly
  Interventions: Drug: 0.12 mg/kg CpG 7909; Drug: Herceptin®
- Cohort 4 (Experimental): 0.16 mg/kg CpG 7909
  Interventions: Drug: 0.16 mg/kg CpG 7909; Drug: Herceptin®

INTERVENTIONS:
Drug: 0.04 mg/kg CpG 7909 — 0.04 mg/kg CpG 7909 by subcutaneous Injection once weekly until progression or 24 weeks
  Other Names: PF-03512676, ProMune
  Arms: Cohort 1
Drug: Herceptin® — Herceptin® (maintenance dose per the manufacturer's directions) followed by a subcutaneous injection of CpG 7909.
  Other Names: Trastuzumab
  Arms: Cohort 1
Drug: 0.08 mg/kg CpG 7909 — 0.08 mg/kg CpG 7909 by subcutaneous Injection once weekly until progression or 24 weeks
  Other Names: PF-03512676, ProMune
  Arms: Cohort 2
Drug: Herceptin® — Herceptin® (maintenance dose per the manufacturer's directions) followed by a subcutaneous injection of CpG 7909.
  Other Names: Trastuzumab
  Arms: Cohort 2
Drug: 0.12 mg/kg CpG 7909 — 0.12 mg/kg CpG 7909 by subcutaneous Injection once weekly until progression or 24 weeks
  Other Names: PF-03512676, ProMune
  Arms: Cohort 3
Drug: Herceptin® — Herceptin® (maintenance dose per the manufacturer's directions) followed by a subcutaneous injection of CpG 7909.
  Other Names: Trastuzumab
  Arms: Cohort 3
Drug: 0.16 mg/kg CpG 7909 — 0.16 mg/kg CpG 7909 by subcutaneous Injection once weekly until progression or 24 weeks
  Other Names: PF-03512676, ProMune
  Arms: Cohort 4
Drug: Herceptin® — Herceptin® (maintenance dose per the manufacturer's directions) followed by a subcutaneous injection of CpG 7909.
  Other Names: Trastuzumab
  Arms: Cohort 4

SUMMARY:
To determine the safety and efficacy of CPG 7909 Injection given with Herceptin to patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer with metastases
* Tumor that has overexpression of HER2 as documented by being either FISH-positive or HER2/neu 3+ confirmed by immunohistochemistry
* Patients may have had up to three prior chemotherapy regimens for metastatic disease, which may have been given in combination with Herceptin® and which may have been discontinued due to toxicities. In addition, patients may have had adjuvant chemotherapy.
* Phase II only: Must have measurable disease by RECIST criteria (defined in section 8) with at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques, or as > 10 mm with spiral CT scan

Exclusion Criteria:

* Any prior therapy with anthracycline + Herceptin® concurrently
* Significant cardiovascular disease (e.g., NYHA class 3 congestive heart failure, myocardial infarction within the past 6 months, unstable angina; coronary angioplasty within the past 6 months, uncontrolled atrial or ventricular cardiac arrhythmias) or left ventricular ejection fraction < 50%
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Phase I: To evaluate the safety and tolerability of several dose levels of CPG 7909 (up to a maximum of 0.16 mg/kg) and to determine the maximum tolerated dose (MTD)* of CPG 7909 in combination with Herceptin® | 24 weeks
Phase II: To evaluate tumor response and safety of CPG 7909 (at the MTD as determined in Phase I) in combination with Herceptin® in patients with metastatic breast cancer. | 24 weeks

SECONDARY OUTCOMES:
Phase I To evaluate tumor response, duration of response, time to disease progression, ECOG performance status, and survival time. | 24 weeks
Phase II To evaluate duration of response, time to disease progression, ECOG performance status, and survival time. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Berkely, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Dearborn, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, West Bloomfield, Michigan
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Burlington, Vermont

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C015&StudyName=CPG%207909%20Plus%20Herceptin%AE%20In%20Patients%20With%20Metastatic%20Breast%20Cancer